CLINICAL TRIAL: NCT04493515
Title: Oral Oxytocin's Effects on Attention Control: An Eye-tracking Study
Brief Title: Oral Oxytocin's Effects on Attention Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-69
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Healthy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Between-subject randomized placebo-controlled double-blind pharmacological eye-tracking design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Oxytocin (Experimental): Oxytocin orally (24 IU)
  Interventions: Drug: Oral Oxytocin
- Oral Placebo (Placebo Comparator): Placebo orally (24 IU, identical ingredients, except the active agent)
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral Oxytocin — Administration of oxytocin orally (24 IU)
  Arms: Oral Oxytocin
Drug: Oral Placebo — Administration of placebo orally (24 IU)
  Arms: Oral Placebo

SUMMARY:
The main aim of the study is to investigate whether orally administered oxytocin (24IU) could modulate attention control using a social-emotional saccade/antisaccade eye-tracking paradigm.

DETAILED DESCRIPTION:
Numerous studies have reported the effect of intranasally administered oxytocin on attentional processing including stimulus-driven bottom-up processing and top-down goal-directed inhibitory control. However, it is unclear whether the functional effects are mediated by the peptide directly entering the brain or indirectly via raising peripheral concentrations. One possible method of producing a similar pattern of increased peripheral oxytocin concentrations but without the possibility of direct entry into the brain would be to administer the peptide lingually. In the present double-blind, between-subject, placebo-controlled study, 80 healthy male subjects will be recruited and receive either oxytocin (24IU) or placebo control administered orally (lingual). 45 minutes after treatment subjects are required to complete a social-emotional saccade/antisaccade eye-tracking paradigm. This paradigm uses social (happy, sad, angry, fear, and neutral faces) as well as non-social (oval shapes) stimuli to explore social- and emotion-specific effects of orally administered oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy participants
* Non smokers

Exclusion Criteria:

* Previous or current medical, psychiatric, neurological disorder
* Regular medication
* Use of any psychoactive substances in the 24 hours before experiment
* Contra-indications for oxytocin
* Contra-indications for eye-tracking data acquisition

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of oral oxytocin administration on saccade/antisaccade latencies towards social (facial) versus non-social (shape) stimuli | 45 minutes - 100 minutes after treatment
  Comparison between social-specific saccade/antisaccade latencies (in milliseconds) between the oxytocin and placebo treatment conditions
Effect of oral oxytocin administration on error rates of saccade/antisaccade for social (facial) versus non-social (shape) stimuli | 45 minutes - 100 minutes after treatment
  Comparison between social-specific error rates of saccade/antisaccade between the oxytocin and placebo treatment conditions.

SECONDARY OUTCOMES:
Emotion-specific effects of oral oxytocin administration on saccade/antisaccade latencies towards the separate facial emotions | 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade latencies (in milliseconds) between the oxytocin and placebo treatment conditions
Emotion-specific effects of oral oxytocin administration on saccade/antisaccade error rates for the separate facial emotions | 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade error rates between the oxytocin and placebo treatment conditions

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China (UESTC)
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No